CLINICAL TRIAL: NCT03332563
Title: Web-based Self-management of Adolescent Chronic Pain: National Implementation Project
Brief Title: WebMAP Mobile Self-management of Adolescent Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Connecticut Children's Medical Center (Other); Children's Mercy Hospital Kansas City (Other); C.S. Mott Children's Hospital (Other); Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Tonya Palermo, Professor, Anesthesiology and Pain Medicine, Seattle Children's Hospital
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: Pfizer 27971161
Record Dates: First submitted 2017-10-29; First posted 2017-11-06 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Chronic Pain
Keywords: Adolescent; Cognitive Behavioral Therapy; Chronic Pain; smartphone application; internet-delivered
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: This study will employ a stepped wedge cluster randomized design in which clinic sites are randomized sequentially to initiate the intervention. Prior to initiating patient recruitment, each of the 8 clinics will be randomized to one of two waves in the stepped wedge design. During the non-exposure periods, patients will receive usual care from the clinic.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WebMAP Mobile (Experimental): Adolescent participants assigned to this arm will receive access to the WebMAP mobile program delivering cognitive-behavioral intervention for chronic pain. Parents of adolescents will receive access to cognitive-behavioral strategies for parents on the WebMAP parent web site.
  Interventions: Behavioral: Cognitive-behavioral intervention for chronic pain
- Usual care (No Intervention): Participants assigned to this arm will receive usual care from the pain or specialty clinic during the non-exposure periods in the stepped wedge design.

INTERVENTIONS:
Behavioral: Cognitive-behavioral intervention for chronic pain — WebMAP is a technology-based cognitive-behavioral intervention program that teaches relaxation skills, pain coping strategies and parent behavioral and communication techniques to youth with chronic pain and their parents.
  Arms: WebMAP Mobile

SUMMARY:
Approximately 5-8% of children report severe chronic pain and disability. Although evidence supports pain-self management as effective for reducing pain and disability, data show that most youth do not have access to this intervention. The investigative team's prior studies demonstrate that technology-delivered pain self-management (WebMAP program) can reduce barriers to care, is feasible, acceptable, and effective in reducing pain-related disability and improving anxiety and depression in youth with chronic pain. In this trial, the investigators propose an implementation project to address critical challenges in nationwide dissemination of the WebMAP pain self-management program. Using a hybrid effectiveness-implementation trial design, 8 clinics from across the U.S. will participate in a pragmatic randomized controlled trial with a stepped wedge design to sequentially implement WebMAP in the clinics following randomized usual care periods. Data will be collected from clinic records, web and app administrative tracking, and provider surveys to gather information on adoption and implementation following the Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM) public health impact framework. Individual patient-level pain outcomes will be collected from 140 patients to evaluate intervention effectiveness. The expected outcome of the project is to yield a strategic approach for a nationwide technology-delivered pain self-management intervention for youth with chronic pain that can be readily sustained in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

1. child age 10-17 years,
2. has chronic pain defined as pain present for at least 3 months, and
3. has access to a smartphone or web-enabled device (e.g., laptop, computer, iPad).

Exclusion Criteria:

1. non-English speaking,
2. presently in a psychiatric crisis,
3. cognitive impairments or intellectual disabilities (has to be able to complete surveys independently),
4. does not have access to a smartphone, computer, or internet, and
5. is unable to read at the 5th grade level.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 143 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Change in activity limitations | Baseline to 3 month followup
  The 9-item Child Activity Limitations Interview (CALI-9) will be completed on the online diary to rate perceived difficulty in completing 9 daily activities due to pain

SECONDARY OUTCOMES:
Change in pain intensity | Baseline to 3 month followup
  Pain intensity will be measured prospectively on the 11-point Pain Numeric Rating Scale (NRS) with anchors of 0 (no pain) to 10 (worst pain possible). Average scores over 7-day assessment periods will be used in analyses.
Change in anxiety and depressive symptoms | Baseline to 3 month followup
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Emotional Distress scale is an 8-item scale of anxiety with scores ranging from 8 to 40 (higher scores indicate greater fear, anxious misery, and hyperarousal). The 8-item scale of depressive symptoms has scores ranging from 8 to 40 with higher scores indicating greater depressive symptoms. Total anxiety and total depression T-scores will be used in analyses.
Change in pain-efficacy | Baseline to 3 month followup
  Pain Self-Efficacy Scale-4 is a 4-item measure that assesses beliefs in carrying out activities when in pain. Total sum score ranging from 0 to 24 will be used in analysis with higher scores representing greater self-efficacy.
Patient's global impression of change | 3 month followup
  1-item measure asking about change since receiving treatment
Change in parent behavior | Baseline to 3 month followup
  Parents report on their protective behaviors on the Adult Responses to Child Symptoms (ARCS), a 29-item scale with subscale scores for three factors, Protect, Minimize, Distract and Monitor. Each subscale is scored by computing the mean of the item responses ranging from 0 to 4 (higher scores indicate more maladaptive behaviors)
Change in parent emotional distress | Baseline to 3 month followup
  Parents report on their anxiety and depression symptoms on the PROMIS Adult Emotional Distress scale. This includes a 4-item scale of anxiety with scores ranging from 4 to 20 (higher scores indicate greater anxiety), and a 4-item scale of depression with scores ranging from 4 to 20 (higher scores indicate greater depression. Total anxiety and depression scale T-scores will be used in analyses.
Change in insomnia severity | Baseline to 3 month followup
  Insomnia Severity Index is a 7-item self-report measure. A 5-point Likert scale is used to rate each item about the severity and impact of insomnia symptoms with scores ranging from 0 to 28 (higher scores indicate greater insomnia sympotoms). A Total score will be used in analyses.

OTHER OUTCOMES:
Adoption - setting level | Assessed at 24 months
  Proportion of children referred to WebMAP at each clinic/Number seen in each clinic
Reach | Assessed at 24 months
  Number of people agree to participate/Number of eligible participants referred for intervention
Implementation, organization level | Assessed at 24 months
  Provider survey regarding feasibility of implementing WebMAP and attitudes toward adoption
Maintenance, organization level | Assessed at 24 months
  Proportion of clinics agreeing to continue using WebMAP

CONTACTS AND LOCATIONS:
Overall Officials: Tonya Palermo, PhD, Principal Investigator — Seattle Children's Hospital
Locations (5):
- United States (5):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palermo TM, de la Vega R, Dudeney J, Murray C, Law E. Mobile health intervention for self-management of adolescent chronic pain (WebMAP mobile): Protocol for a hybrid effectiveness-implementation cluster randomized controlled trial. Contemp Clin Trials. 2018 Nov;74:55-60. doi: 10.1016/j.cct.2018.10.003. Epub 2018 Oct 2. PMID 30290276